CLINICAL TRIAL: NCT00167427
Title: Genotoxicity Assessment for Patients Receiving Large Field Irradiation
Brief Title: Genotoxicity Assessment for Patients Undergoing Radiation Treatment
Status: Completed | Type: Observational
Sponsor: Yuhchyau Chen (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor-Investigator, Yuhchyau Chen, Investigatory, University of Rochester
Organization: University of Rochester (Other)
Other Study IDs: URCC 3705; 1U19AI067733-01 (NIH)
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the research study is to evaluate an automated, laser-based technique for measuring DNA damage caused by radiation during cancer treatment in immature red blood cells.

DETAILED DESCRIPTION:
Correlative studies: analysis of RT effect on genotoxicity by assessing cytogenetic changes (dicentrics), micronucleated lymphocytes (MN-lymph), and micronucleated reticulocytes (MN-RET) using peripheral blood of patients receiving radiation.

i) document the kinetics by which radiation-induced MN-RET enter the peripheral blood stream.

ii) benchmark the MN-RET endpoint against current gold-standard biodosimetry endpoints-dicentrics and MN-lymphocytes.

iii) measure inter-individual variation in baseline and radiation-induced MN-RET frequencies.

iv) in collaboration with several FCM-equipped laboratories, evaluate the transferability of the human MN-RET scoring assay.

ELIGIBILITY:
Inclusion Criteria:

* Patients that are scheduled to begin radiotherapy to the large-field chest region are eligible if:

  * Daily radiation dose is between 1.8 and 5 Gy/day
  * Any single dimension of field size is ≥ 15 cm
  * Provision of written informed consent

or

* Or patients receiving IMRT or Tomotherapy, when low-dose radiation is spread out to the normal tissues, irrespective of daily radiation doses.
* Or patients receiving radionucleotides as part of the medical treatment (cancer or non-malignant conditions)
* Or patients who will receive diagnostic CT scans, PET/CT scans, mammograms, or diagnostic imaging requiring radionucleotides

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that are scheduled to begin radiotherapy to the large-field chest region
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2006-04; Primary Completion 2024-02-23 (Actual); Study Completion 2024-02-23 (Actual)

PRIMARY OUTCOMES:
Measure the Change in MN-RET in the blood | Baseline and 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Yuhchyau Chen, MD, Ph.D, Principal Investigator — Universtiy of Rochester, Dept of Radiation Oncology
Locations (1):
- University of Rochester, Dept. Radiation Oncology, Rochester, New York, United States